CLINICAL TRIAL: NCT03442361
Title: Olive Oil and Soybean 1 Oil Based Intravenous Lipid Emulsions, Liver Biochemistry and Clinical Outcomes
Brief Title: Olive Oil and Soybean 1 Oil Based Intravenous Lipid Emulsions, Liver Chemistry and Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Maitreyi Raman, Principal Investigator, University of Calgary
Other Study IDs: AJCN Raman
Record Dates: First submitted 2018-01-23; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Parenteral Nutrition Associated Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intralipid: Standard soybean oil-based therapy
- Clinoleic: Olive oil based therapy

SUMMARY:
Background: Intravenous lipid emulsions (IVLE) are an essential component of parenteral nutrition (PN). Omega-6 reducing strategies may improve outcomes, including reduced PN associated liver disease.

Objective: The primary objective was to compare serum alkaline phosphatase (ALP), among surgical and medical patients provided with either Intralipid or Clinoleic lipid emulsions.

Design: In this quasi-experimental study the medical records of surgical and medical adult patients were reviewed from 3 Canadian hospitals that received PN with either soybean oil (Intralipid) or predominantly olive oil (Clinoleic) based lipid emulsions for at least 7 consecutive days.

DETAILED DESCRIPTION:
A few small studies have shown that a predominantly olive oil based IVLE is well tolerated and safe, however the clinical relevance of this IVLE is uncertain as no clear benefit in outcomes has been observed in small randomized clinical trials. Given the limited data available for the adult population reporting on the experience with olive oil based IVLE, we designed a quasi-experimental study to review our experience with Clinoleic compared to Intralipid. The primary objective was to compare the impact of Intralipid and Clinoleic IVLE on serum alkaline phosphatase (ALP), pre-PN to after one week of PN (i.e. between day 8 to 16 post-PN initiation), while controlling for the ordered lipid dosing. Secondary objectives were to assess if there were differences between the IVLEs on the remaining liver function tests, lipid dosing, incidence of infectious complications, length of stay in hospital and 30- day mortality.

This retrospective quasi-experimental chart review was conducted in 3 tertiary care hospitals in Calgary, AB between July 01, 2012 to June 30, 2013 and July 01, 2014 to June 30, 2015. Standard soybean oil-based therapy, Intralipid was the only available IVLE in Calgary, AB until July 2013, at which time predominantly olive oil Clinoleic was approved as an alternative in the hospital formulary, accounting for the dates chosen for the study. Ethics approval from the Conjoint Health Research and Ethics Board at the University of Calgary was obtained prior to the initiation of the study.

ELIGIBILITY:
Inclusion Criteria:

* admitted to hospital who received PN with Intralipid or Clinoleic IVLEs for at least 7 consecutive days.

Exclusion Criteria:

* baseline liver disease
* home PN prior to admission
* ALP and total bilirubin (TB) not available within 3 days prior to PN start as well as between days 8 to 16 post PN start
* receipt of Diprivan 1%® (Propofol 116 - AstraZeneca Canada Inc., Mississauga, Canada) during PN support period
* enteral nutrition providing greater than 600 Kcal daily for longer than half of time period on PN
* oral intake of greater than 50% of hospital meal tray contents for longer than half of the PN support time period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study patients included adult patients (> 18 years) admitted to hospital who received PN with Intralipid or Clinoleic IVLEs for at least 7 consecutive days
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Serum ALP Level | 8 to 16 days after PN initiation
  Difference between Intralipid and Clinoleic groups

SECONDARY OUTCOMES:
Serum ALT | 8 to 16 days after PN initiation
  Difference between Intralipid and Clinoleic groups
Serum GGT | 8 to 16 days after PN initiation
  Difference between Intralipid and Clinoleic groups
Serum TB | 8 to 16 days after PN initiation
  Difference between Intralipid and Clinoleic groups
Serum BD | 8 to 16 days after PN initiation
  Difference between Intralipid and Clinoleic groups
Serum TG | 8 to 16 days after PN initiation
  Difference between Intralipid and Clinoleic groups
IVLE prescriptions dosing | Day 3 to 16 after PN initiation
  Difference between Intralipid and Clinoleic groups
All cause mortality | By 30 days after PN initiation
  Difference between Intralipid and Clinoleic groups
Length of hospital stay | During PN Period
  Difference between Intralipid and Clinoleic groups
Infectious complications incidence | During PN Period
  Difference between Intralipid and Clinoleic groups

CONTACTS AND LOCATIONS:
Overall Officials: Maitreyi Raman, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No